CLINICAL TRIAL: NCT04332913
Title: Efficacy and Safety of Tocilizumab in the Treatment of Patients With Respiratory Distress Syndrome and Cytokine Release Syndrome Secondary to COVID-19: a Proof of Concept Study
Brief Title: Efficacy and Safety of Tocilizumab in the Treatment of SARS-Cov-2 Related Pneumonia
Acronym: TOSCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Prof. Roberto Giacomelli, Full Professor, University of L'Aquila
Other Study IDs: 0064468/20
Record Dates: First submitted 2020-03-26; First posted 2020-04-03 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: COVID-19 Pneumonia
Keywords: Tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The current spread of the COrona VIrus Disease-2019 (COVID-19) epidemic in Italy, and the current lack of effective and approved drugs for its treatment, poses the problem of Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infected patients management, especially those who underwent to experience COVID-19 complications, such as CRS. This unmet need becomes more severe if the investigator consider that, the COVID-19 mortality stands around 2% in the general population, but it rises to 49% when considering intensive care unit (ICU) patients. To increase the chances of survival of these patients, the compassionate use of the available drugs is required, based on literature data, to the best of our abilities. ICU patients with cytokine release syndrome (CRS) secondary to COVID-19, show increased production of pro-inflammatory cytokines, including interleukin (IL-6), IL-2, IL-7, IL-10, tumor necrosis factor (TNF)-α and interferon (INF)γ, similar to that found in patients who develop CRS secondary to Chimeric Antigen Receptor-T (CAR-T) therapy. Although immuno-modulatory therapy is not routinely recommended in COVID-19 pneumonia, tocilizumab might have a rationale in those patients who develop CRS, blocking the complications caused by high levels of IL-6, and possibly preventing the development of a multi-organ failure. Reassuring data in this sense, come from the first studies conducted in China. In a Chinese pilot study, Xiaoling Xu and collaborators used tocilizumab (at a dosage of 400 mg iv in a single dose, with a possible second dose in case of no clinical response) in patients with COVID-19 in the presence of one of the following criteria: i) respiratory rate ≥ 30 acts/min; ii) SpO2 ≤ 93% in ambient air; iii) PaO2/FiO2 ≤ 300 mmHg. In the 21 patients treated with tocilizumab a significant reduction in IL-6 levels and fever, with improvement in lung function, was demonstrated. Besides, 90% of treated patients showed an improvement in the radiological picture, in terms of a decrease in the frosted glass areas, and a return to normal lymphocytes count in the peripheral blood. This is a prospective observational clinical study and it is aimed at verifying tocilizumab efficacy and safety in patients with COVID-19 complicated by acute distress respiratory syndrome (ARDS) and CRS.

ELIGIBILITY:
Inclusion Criteria:

* All gender patients aged ≥ 18 years;
* Patients with SARS-CoV-2 infection confirmed by tests (RT-PCR) and pulmonary involvement, hospitalized, at the end of the initial phase of high viral load of COVID-19 (apyretic> 72 hours and / or at least 7 days after onset of symptoms);
* Worsening of respiratory exchanges such as to require non-invasive or invasive ventilation support (BCRSS score ≥ 3).
* High levels of IL-6 (> 40 pg/mL) or alternatively CRP and/or ferritin and/or D-dimer and/or fibrinogen values higher than the reference values or rapidly increasing;
* Signature of informed consent.

Exclusion Criteria:

* Alanine aminotransferase and/or Aspartate aminotransferase (ALT / AST) > 5 times compared to normal laboratory values.
* Presence of a chronic renal failure ≥ 4 stage (glomerular filtrate values <30 ml/min/1.73 m2).
* Presence of neutropenia (neutrophils count < 500 / mm3).
* Platelet count less than 50 x 103/μL.
* Documented sepsis from other pathogens other than SARS-CoV-2.
* Presence of co-morbidities associated, in clinical judgment, with an unfavourable outcome.
* Complicated diverticulitis and / or intestinal perforation.
* Skin infection in progress (e.g. dermohypodermitis not controlled by antibiotic therapy).
* Immuno-suppressive anti-rejection therapy.
* Pregnancy or woman of childbearing age who does not use contraceptive and/or breastfeeding measures.
* Previous ischemic attack or myocardial infarction.
* NYHA class III or IV heart failure.
* Severe depressive syndrome or other psychiatric disease which, in the opinion of the doctor, can preclude patient participation in the study.
* Presence of known malignant neoplasms.
* Clinically significant history of alcohol abuse or drug addiction which, in the opinion of the doctor, may preclude the subject's participation in the study.
* Any condition which, in the opinion of the doctor, precludes the possibility of using the study drug provided for in the RCP.
* Any other laboratory condition or parameter that, in the doctor's judgment, precludes the subject's participation in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients with pneumonia requiring hospitalization
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete recovery defined as fever disappearance and return to normal peripheral oxygen saturation values (SpO2) after 14 days from the end of treatment with tocilizumab. | 14 days
  Fever normalization criteria: Temperature <36.6 ° C for at least 72 hours; SpO2 normalization criterion: SpO2> 94% for at least 72 hours

SECONDARY OUTCOMES:
Percentage of patients achieving a score <3 on the Brescia-COVID respiratory severity scale (BCRSS) after the last tocilizumab administration. | 24 hours
Percentage of patients with partial recovery defined as the disappearance of fever 14 days after the end of treatment with tocilizumab. | 14 days
  Fever normalization criteria: Temperature <36.6 ° C for at least 72 hours
Duration of hospitalization | 14 days
  days
Time to the first negative SARS-CoV-2 negative RT-PCR test | 14 days
  days
Changes from the baseline in the white blood cell count | 7, 14 days
  number/microliter
Changes from the baseline in the lymphocyte populations (cluster of differentiation (CD)3+CD4+, CD3+CD8+, CD19+, Th17) | 7, 14 days
  number/microliter
Changes from the baseline of c-reactive protein (CRP) values | 7, 14 days
Changes from the baseline of Ferritin values | 7, 14 days
Changes from the baseline of BNP values | 7,14 days
Changes from the baseline of CK-MB values | 7,14 days
Changes from the baseline of Troponin values | 7,14 days
Changes from the baseline of LDH values | 7,14 days
Changes from the baseline of myoglobulin values | 7,14 days
Changes in myocardial ischemia signs at the electrocardiographic trace (YES or NO) | 7,14 days
  (ST segments elevation or depression, T-wave changes)
Rate of adverse events report during and after tocilizumab | 14 days
Mortality (number of Partecipants, cause and timing) | 12 weeks
Percentage of patients who develop autoimmune diseases | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Salvatore, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Hays P, Costello C, Asudani D. Clinical care of chimeric antigen receptor T-cell patients and managing immune-related adverse effects in the ambulatory and hospitalized setting: a review. Future Oncol. 2019 Dec;15(36):4235-4246. doi: 10.2217/fon-2019-0467. Epub 2019 Nov 27. PMID 31773980
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Hunter CA, Jones SA. IL-6 as a keystone cytokine in health and disease. Nat Immunol. 2015 May;16(5):448-57. doi: 10.1038/ni.3153. PMID 25898198
- [Background] Le RQ, Li L, Yuan W, Shord SS, Nie L, Habtemariam BA, Przepiorka D, Farrell AT, Pazdur R. FDA Approval Summary: Tocilizumab for Treatment of Chimeric Antigen Receptor T Cell-Induced Severe or Life-Threatening Cytokine Release Syndrome. Oncologist. 2018 Aug;23(8):943-947. doi: 10.1634/theoncologist.2018-0028. Epub 2018 Apr 5. PMID 29622697
- [Background] Pathan N, Hemingway CA, Alizadeh AA, Stephens AC, Boldrick JC, Oragui EE, McCabe C, Welch SB, Whitney A, O'Gara P, Nadel S, Relman DA, Harding SE, Levin M. Role of interleukin 6 in myocardial dysfunction of meningococcal septic shock. Lancet. 2004 Jan 17;363(9404):203-9. doi: 10.1016/S0140-6736(03)15326-3. PMID 14738793
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Salehi S, Abedi A, Balakrishnan S, Gholamrezanezhad A. Coronavirus Disease 2019 (COVID-19): A Systematic Review of Imaging Findings in 919 Patients. AJR Am J Roentgenol. 2020 Jul;215(1):87-93. doi: 10.2214/AJR.20.23034. Epub 2020 Mar 14. PMID 32174129
- [Background] Shimabukuro-Vornhagen A, Godel P, Subklewe M, Stemmler HJ, Schlosser HA, Schlaak M, Kochanek M, Boll B, von Bergwelt-Baildon MS. Cytokine release syndrome. J Immunother Cancer. 2018 Jun 15;6(1):56. doi: 10.1186/s40425-018-0343-9. PMID 29907163
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] van der Stegen SJ, Davies DM, Wilkie S, Foster J, Sosabowski JK, Burnet J, Whilding LM, Petrovic RM, Ghaem-Maghami S, Mather S, Jeannon JP, Parente-Pereira AC, Maher J. Preclinical in vivo modeling of cytokine release syndrome induced by ErbB-retargeted human T cells: identifying a window of therapeutic opportunity? J Immunol. 2013 Nov 1;191(9):4589-98. doi: 10.4049/jimmunol.1301523. Epub 2013 Sep 23. PMID 24062490
- [Background] Winkler U, Jensen M, Manzke O, Schulz H, Diehl V, Engert A. Cytokine-release syndrome in patients with B-cell chronic lymphocytic leukemia and high lymphocyte counts after treatment with an anti-CD20 monoclonal antibody (rituximab, IDEC-C2B8). Blood. 1999 Oct 1;94(7):2217-24. PMID 10498591
- [Background] Xu X, Han M, Li T, Sun W, Wang D, Fu B, Zhou Y, Zheng X, Yang Y, Li X, Zhang X, Pan A, Wei H. Effective treatment of severe COVID-19 patients with tocilizumab. Proc Natl Acad Sci U S A. 2020 May 19;117(20):10970-10975. doi: 10.1073/pnas.2005615117. Epub 2020 Apr 29. PMID 32350134
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Result] Gorbalenya AE, Baker SC, Baric RS, et al. Severe acute respiratory syndrome-related coronavirus: The species and its viruses - a statement of the Coronavirus Study Group. BioRxivchinaXiv:202003.00026v172020:2020.02.07.937862.